CLINICAL TRIAL: NCT06067412
Title: Efficacy of Phenytoin vs Levetiracetam in Status Epilepticus at Institute of Child Health,Faisalabad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Ali Raza Chaudhry, Senior Registrar Paediatric Surgery, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 184-86
Record Dates: First submitted 2023-09-10; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Status Epilepticus
Keywords: Efficacy; Phenytoin; Levetiracetam
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam; Phenytoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- levetiracetam (Active Comparator): levetiracetam at a dose of 30 mg/kg diluted in 50 ml of normal saline in 15 minutes followed by a maintenance dose of 30mg/kg/day divided in two doses 12 hours apart after initial loading dose.
  if seizures recurred after the first loading dose an additional 10mg/kg of the same drug was given over 10 minutes. If seizures recurred, the patients were loaded with sodium valporate 30 mg/kg diluted in 50 ml normal saline in 15 minutes.
  Interventions: Drug: Levetiracetam
- phenytoin (Active Comparator): I/V phenytoin at 20 mg/kg diluted in 50ml normal saline in 15 minutes followed by maintenance dose of 5 mg/kg/day divided in two doses 12 hours apart.
  if seizures recurred after the first loading dose an additional 10mg/kg of the same drug was given over 10 minutes. If seizures recurred, the patients were loaded with sodium valporate 30 mg/kg diluted in 50 ml normal saline in 15 minutes.
  Interventions: Drug: Phenytoin

INTERVENTIONS:
Drug: Levetiracetam — Efficacy in fits
  Arms: levetiracetam
Drug: Phenytoin — Efficacy in fits
  Arms: phenytoin

SUMMARY:
Status epilepticus is the second most common neurologic emergency in children. Morbidity and mortality are considerable; thus, timely termination of convulsive status epilepticus is the primary goal of management to avoid these risks Our objective was to compare the efficacy of phenytoin and Levetiracetam in status epilepticus in children.

This study was done in the pediatric emergency department of Children Hospital Faisalabad.

A total of 70 patients were randomly allocated to one of the groups by a computer-generated random number table according to their admission in an emergency. Children in group A were given levetiracetam. Children in group B were given I/V phenytoin. For both groups if seizures recurred after the first loading dose an additional 10mg/kg of the same drug was given over 10 minutes.

The patients were monitored to see whether there was any recurrence of seizure activity in the subsequent 24 hours. Seizure control was defined as the absence of seizure within 24 hours after the initial loading of the drug.

DETAILED DESCRIPTION:
OPERATIONAL DEFINITION

Status Epilepticus:

It is defined as continuous seizure activity or recurrent seizure activity without regaining of consciousness lasting for more than 5 minutes.

Efficacy:

Efficacy means control of seizures without supplemental aid of either medication or no recurrence with in twenty-four hours.

HYPOTHESIS H0: There is no significant difference between efficacy of Phenytoin and Levetiracetam in Status Epilepticus in Children H1: There is significant difference between efficacy of Phenytoin and Levetiracetam in Status Epilepticus in Children.

MATERIAL AND METHODS

STUDY DESIGN:

Randomized Controlled Trial (RCT). SETTING This study was done in pediatric emergency department of Children Hospital Faisalabad.

DURATION OF STUDY The duration of study was six months after the approval of synopsis From: 1/8/2022 to 31/1/2023

SAMPLE SIZE:

By using WHO sample size calculator for two proportions:

p1=96%7, p2=59.6%7 power of study = 90% Level of significance = 5% Sample Size = 70 (35 in each group) SAMPLING TECHNIQUE Nonprobability consecutive sampling

DATA COLLECTION PROCEDURE After approval from IRB, patient fulfilling the inclusion criteria were enrolled. Written informed consent was taken and data was collected through predesigned Performa in emergency of Children Hospital Faisalabad. The patients were randomly allocated to one of the group by computer generated random number table according to their admission in emergency. After taking full care of Airway and Breathing I/V line was established children who presented with active seizures were given Diazepam at a dose of 0.1 mg /kg I/V slowly stat followed by I/V levetiracetam or phenytoin according to group allocation. Children with recent history of status epilepticus but now present with no active seizures were given only I/V levetiracetam or phenytoin.

Children in group A was given levetiracetam at a dose of 30 mg/kg diluted in 50 ml of normal saline in 15 minutes followed by a maintenance dose of 30mg/kg/day divided in two doses 12 hours apart after initial loading dose. Children in group B was given I/V phenytoin at 20 mg/kg diluted in 50ml normal saline in 15 minutes followed by maintenance dose of 5 mg/kg/day divided in two doses 12 hours apart. For both groups if seizures recurred after the first loading dose an additional 10mg/kg of the same drug was given over 10 minutes. If seizures recurred, the patients were loaded with sodium valporate 30 mg/kg diluted in 50 ml normal saline in 15 minutes.

The parameters which include level of consciousness (GCS), heart rate, respiratory rate, blood pressure and oxygen saturation was noted first at the time of admission and then again at 30 minutes, 1hour, 6hour, 12hour and 24 hours. The patients were monitored to see whether there was any recurrence of seizure activity in subsequent 24 hours. Seizure control was defined as the absence of seizure for 24 hours after the initial loading of the drug.

DATA ANALYSIS PROCEDURE:

Data was analyzed by SPSS V-25. Frequency and Percentage was calculated for all qualitative variables like gender, type of seizures and efficacy. Mean ± Standard Deviation was calculated for all quantitative variables like age and weight. Efficacy was compared by applying chi-square test between two groups. Effect modifiers like age, gender, weight and type of seizures were controlled by stratification. Post stratification chi-square test was applied P ≤ 0.05 was taken as significant.

DISCUSSION In order to avoid neurologic and systemic disease, effective treatment of status epilepticus is necessary. The prompt identification and complete cessation of seizures have to be the overarching objectives of any therapy. In order for an anticonvulsant medication to be successful in treating status epilepticus, it must be given intravenously. This allows for the medication to be delivered to the brain more quickly while also reducing the likelihood of major side effects on the nervous system. There is more than one medication available, and each one has its own set of benefits and drawbacks.

There have been a number of studies published on the efficacy of both drugs but the data showing the relative effect of both drugs is still insufficient. In Pakistan there were only few researches showing efficacy of both drugs, this leads to the thought to conduct this particular research in our hospital to compare their relative efficacy in order to improve the seizure control time in our hospital and benefit patients with the best available drug.

Many randomized clinical trials clearly supports the use of benzodiazepine as the first line treatment in status epilepticus.But, if the seizure control was not established than 2nd line drugs phenytoin , levetiracetam and sodium valporate were used.There were mixed results in terms of efficacies of both drugs .In one study, mean age was 4.09 years with male predominance and most common type of seizures were generalized tonic clonic (74%).The seizure control time in all 104 patients was within 40 minutes. Seizures were better controlled in group 1 (levetiracetam 96%) as compared to group 2 (phenytoin 59.6%) in 1st 24 hours (P=0.0001).

Numerous studies have shown that levetiracetam is a safer AED to give than phenytoin, despite the fact that both medications are as effective in treating SE. This is the case despite the fact that the two drugs have equivalent efficacies. The incidence of adverse effects associated with the therapy with phenytoin was considerably higher than the incidence of adverse effects associated with levetiracetam. The most prevalent adverse event was acute hypotension.

When treating SE, another clinical investigation found that intravenous (IV) fosphenytoin was linked with much more vasopressor use than levetiracetam. This was mostly owing to the hypotension that was generated by the treatment.The danger of hypotension that is linked with intravenous (IV) phenytoin and fosphenytoin might contribute to worse patient outcomes. This is because maintaining cerebral blood perfusion is essential for helping to avoid neuronal impairment in In addition, clinical trials have shown that administering phenytoin intravenously might result in potentially deadly arrhythmias in the heart. Although at first it was believed that phenytoin would lower the risk of cardiac toxicity, it now seems that fosphenytoin also causes cardiac arrhythmias. On the other hand, levetiracetam has a less severe adverse effect profile and shows signs of being well tolerated in a variety of patient demographics when it comes to the treatment of SE.

In comparison to phenytoin, the pharmacokinetics of levetiracetam are more favorable, and it is easier to administer. These are two of the many benefits of utilizing levetiracetam to treat SE.Levetiracetam, in contrast to phenytoin, is not metabolized by the CYP450 enzyme system in the liver. As a result, the likelihood of levetiracetam interacting negatively with other medications that are processed by CYP450 is significantly reduced.

In addition, levetiracetam has a bioavailability that is close to one hundred percent and, in contrast to phenytoin, it does not need to have its dosage closely monitored all the time. Another benefit of levetiracetam is that it has linear pharmacokinetics and a wide therapeutic index, both of which significantly lessen the likelihood that the medication would cause adverse effects. It is essential to note that the administration of levetiracetam is noticeably simpler and more expedient than that of phenytoin. In point of fact, administering a loading dosage of intravenous phenytoin to a patient is a process that is laborious and time-consuming, which further raises the potential for unintended side effects.

The effectiveness of the two medications in treating SE may be comparable; however, levetiracetam is the antiepileptic drug (AED) that is safer and more well tolerated. As a result, it ought to take the place of phenytoin and fosphenytoin for the purpose of ending seizure activity in individuals who are resistant to benzodiazepines.

ELIGIBILITY:
Inclusion Criteria

* Children with status Epilepticus i.e with continuous seizure of 5 min or more or two or more discrete seizures in which there is incomplete recovery of consciousness was included in this study.
* Convulsive states epilepticus,
* Generalized tonic clonic seizures,
* Focal tonic clonic seizures are included.
* Age:6 months to 12 years.
* Gender: Both genders.

Exclusion Criteria:

* Participants on any antiepileptic drug (AED) or having allergic reaction towards phenytoin or Levetiracetam were excluded from the study.
* Non convulsive status epilepticus,
* Absence status epilepticus,
* Myoclonic status epilepticus were excluded.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of phenytoin and Levetiracetam in status epilepticus in children. | Six months whole data was collected who were coming in the emergency department
  The patients were monitored to see whether there was any recurrence of seizure activity in subsequent 24 hours. Seizure control was defined as the absence of seizure for 24 hours after the initial loading of the drug.
To compare the efficacy of phenytoin and Levetiracetam in status epilepticus in children. | Six months
  Others parameters which include level of consciousness (GCS), heart rate in Bpm, respiratory rate per minute, blood pressure with sphygnomanometer and oxygen saturation with pulse oximeter was noted first at the time of admission and then again at 30 minutes, 1hour, 6hour, 12hour and 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hopsital Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No